CLINICAL TRIAL: NCT06383663
Title: A Prospective Multicenter Randomized Controlled Trial of the Prognostic Effects of Supraclavicular Lymph Node Dissection vs. No-dissection in Ipsilateral Supraclavicular Lymph Node Metastasis in Breast Cancer
Brief Title: Supraclavicular Lymph Node Dissection for Ipsilateral Supraclavicular Lymph Node Metastatic Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Weidong Wei, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 308-2019-04-01
Record Dates: First submitted 2024-04-21; First posted 2024-04-25 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer; Ipsilateral Supraclavicular Lymph Node Metastasis
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Supraclavicular lymph node dissection combined with radiotherapy versus radiotherapy alone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supraclavicular lymph node dissection combined with radiotherapy (Experimental): Breast cancer patients with ipsilateral supraclavicular lymph node metastases receive standard radiotherapy after supraclavicular lymph node dissection.
  Interventions: Procedure: Supraclavicular lymph node dissection combined with radiotherapy
- radiotherapy (Placebo Comparator): Breast cancer patients with ipsilateral supraclavicular lymph node metastases receive only standard radiotherapy.
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Procedure: Supraclavicular lymph node dissection combined with radiotherapy — Breast cancer patients in the expreimental cohort with only ipsilateral supraclavicular lymph node metastasis were first treated with supraclavicular lymph node dissection and received standard radiotherapy after surgery.
  Arms: Supraclavicular lymph node dissection combined with radiotherapy
Radiation: radiotherapy — Patients in the control group received only standard radiation therapy.
  Arms: radiotherapy

SUMMARY:
The purpose of this study was to compare the efficacy of surgical dissection of supraclavicular lymph nodes combined with radiotherapy versus radiotherapy alone in patients with ipsilateral supraclavicular lymph node metastasis.

DETAILED DESCRIPTION:
In this study, patients with ipsilateral supraclavicular lymph node positive breast cancer were selected as research subjects. Randomized controlled method was used to study the effects of surgical dissection of supraclavicular lymph node combined with radiotherapy and radiotherapy alone on progression-free survival and overall survival of breast cancer. This RCT aims to explore the best treatment method for ipsilateral supraclavicular lymph node metastasis and to provide the basis for guiding the precise treatment of supraclavicular lymph node chain.

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated primary breast cancer with supraclavicular lymph node metastasis or supraclavicular lymph node metastasis without other metastasis within 5 years after combined therapy; The diagnostic criteria refer to the diagnostic criteria for "primary breast cancer" and "Stage pN3c" in the AJCC Guidelines published on November 8, 2018;
2. Supraclavicular lymph node metastasis was confirmed by pathology;
3. Consent to receive biopsy of breast cancer and supraclavicular lymph node tissue;
4. Patients with primary breast cancer have no history of malignant tumors and have not received chemotherapy, radiotherapy or endocrine therapy;
5. Have at least one measurable target lesion according to RECIST criteria;
6. ECOG score ≦ 1;
7. The level of organ function must meet the following requirements: adequate bone marrow reserve: absolute counts of neutrophils (lobed and band neutrophils) ≥ 1.5×109/L, platelets ≥ 100×109/L, and hemoglobin ≥ 9 g/dL. Liver: Bilirubin <1.5 times the upper limit of normal, alkaline phosphatase (AP), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <3.0 times the upper limit of normal. Renal: Creatinine clearance ≥ 45 mL/min;
8. No distant metastases were found in preoperative imaging examination of whole abdominal color ultrasound, chest CT or MRI, bone scan, or PET/CT;
9. normal mind, can cooperate to complete the treatment;
10. Expected survival ≥36 months
11. In accordance with the requirements of the Ethics Committee, there is an informed consent signed by the patient or her legal representative, or an informed consent signed by the patient and her family.

Exclusion Criteria:

1. The range of metastasis exceeds the neck IV and VB region;
2. En-bloc resection cannot be achieved;
3. Patients with heart, lung, vascular and other diseases cannot receive antitumor therapy;
4. Preoperative examination found distant metastasis;
5. Pregnant, lactating or inflammatory breast cancer patients;
6. Diseases associated with immune, endocrine or cardiovascular systems;
7. Previous history of other tumors or combined with other tumors;
8. Refusing to comply with the study protocol and refusing to sign the informed consent

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
DFS | 5-year
  Disease-free survival

SECONDARY OUTCOMES:
PFS | 3-year
  Progression-free survival
OS | 5-year
  Overall survival

OTHER OUTCOMES:
pCR rate | 1-year
  Pathological complete response rate

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Wei, Professor, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Recht A, Gray R, Davidson NE, Fowble BL, Solin LJ, Cummings FJ, Falkson G, Falkson HC, Taylor SG 4th, Tormey DC. Locoregional failure 10 years after mastectomy and adjuvant chemotherapy with or without tamoxifen without irradiation: experience of the Eastern Cooperative Oncology Group. J Clin Oncol. 1999 Jun;17(6):1689-700. doi: 10.1200/JCO.1999.17.6.1689. PMID 10561205
- [Background] Chen SC, Chen MF, Hwang TL, Chao TC, Lo YF, Hsueh S, Chang JT, Leung WM. Prediction of supraclavicular lymph node metastasis in breast carcinoma. Int J Radiat Oncol Biol Phys. 2002 Mar 1;52(3):614-9. doi: 10.1016/s0360-3016(01)02680-3. PMID 11849781
- [Background] Chang XZ, Yin J, Sun J, Zhang XH, Cao XC. A retrospective study of different local treatments in breast cancer patients with synchronous ipsilateral supraclavicular lymph node metastasis. J Cancer Res Ther. 2013 Nov;9 Suppl:S158-61. doi: 10.4103/0973-1482.122514. PMID 24516053
- [Background] Jung J, Kim SS, Ahn SD, Lee SW, Ahn SH, Son BH, Lee JW, Choi EK. Treatment Outcome of Breast Cancer with Pathologically Proven Synchronous Ipsilateral Supraclavicular Lymph Node Metastases. J Breast Cancer. 2015 Jun;18(2):167-72. doi: 10.4048/jbc.2015.18.2.167. Epub 2015 Jun 26. PMID 26155293
- [Background] Lakatos E. Designing complex group sequential survival trials. Stat Med. 2002 Jul 30;21(14):1969-89. doi: 10.1002/sim.1193. PMID 12111882